CLINICAL TRIAL: NCT03615911
Title: An Open, Single Center Phase I Trial to Assess the Safety, Tolerability and Immunogenicity of Two Ascending Doses of the Candidate Vaccine MVA-MERS-S
Brief Title: Safety, Tolerability and Immunogenicity of Vaccine Candidate MVA-MERS-S
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Marylyn Addo (Other)
Collaborators: Philipps University Marburg (Other); Ludwig-Maximilians - University of Munich (Other); Charite University, Berlin, Germany (Other); Bernhard Nocht Institute for Tropical Medicine (Other Government); University of Cologne (Other)
Responsible Party: Sponsor-Investigator, Marylyn Addo, Prof. Dr. med. Marylyn M. Addo, Principal Investigator, Head of the Department of Infectious Diseases, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UKE-DZIF1-MVA-MERS-S
Record Dates: First submitted 2018-07-20; First posted 2018-08-06 (Actual); Results first posted 2020-10-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: MERS (Middle East Respiratory Syndrome)
Keywords: vaccine; clinical phase 1; modified vaccinia Ankara vector; MERS-CoV
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccination with 10^7 PFU MVA-MERS-S (Experimental): Vaccinations occur on days 0 and 28
  A subgroup will additionally receive a late booster immunization with 10^8 PFU MVA-MERS-S 12 months (+/- 4 months) after prime immunization.
  Interventions: Biological: vaccine candidate MVA-MERS-S
- Vaccination with 10^8 PFU MVA-MERS-S (Experimental): Vaccinations occur on days 0 and 28
  A subgroup will additionally receive a late booster immunization with 10^8 PFU MVA-MERS-S 12 months (+/- 4 months) after prime immunization.
  Interventions: Biological: vaccine candidate MVA-MERS-S

INTERVENTIONS:
Biological: vaccine candidate MVA-MERS-S — vaccination with MVA-MERS-S in two escalating dose regimes

SUMMARY:
The Middle East Respiratory Syndrome Coronavirus (MERS-CoV) is a potentially fatal disease with a reported lethality of up to 40% that is under tight epidemiologic control by the World Health Organization (WHO) and currently without registered prevention or treatment option.

In this phase I first-in-human clinical trial, healthy volunteers in two different dose cohorts will be vaccinated twice with the candidate vaccine MVA-MERS-S. A subgroup will additionally receive a late booster vaccination.

The aim of the study is to assess the safety and tolerability of the candidate vaccine and to characterize its immunogenicity.

DETAILED DESCRIPTION:
The vaccine contains a Modified Vaccinia Virus Ankara (MVA) vector expressing the MERS-CoV spike glycoprotein (S). A total of 24 participants will receive the following vaccine regime:

12 participants will receive 10^7 plaque-forming units (PFU) of MVA-MERS-S on days 0 and 28.

12 participants will receive 10^8 PFU of MVA-MERS-S on days 0 and 28.

Safety and immunogenicity data will be collected throughout the study, which concludes at day 180.

Update March 2019: A subgroup of participants from both dose cohorts will receive a late booster immunization of 10^8 PFU MVA-MERS-S 12 months (+/- 4 months) after prime immunization.

ELIGIBILITY:
Inclusion Criteria:

The participant must not be enrolled before all inclusion criteria (including test results) are confirmed. Subjects meeting all of the criteria listed below will be included in the study:

1. Ability to understand the subject information and to personally sign and date the informed consent to participate in the study, before completing any study related procedures.
2. Provided written informed consent.
3. Healthy male and female participants aged 18 - 55 years inclusive at the time of consent. The date of signing informed consent is defined as the beginning of the screening period. This inclusion criterion will only be assessed at the first screening visit.
4. No clinically significant health problems as determined during medical history and physical examination at screening visit.
5. Body weight in defined relation to height. Body mass index 18.5 - 30.0 kg/m2 and weight >50 kg at screening.
6. Females of child-bearing potential who agree to apply effective contraception methods (defined as a contraceptive method with failure rate of less than 1% per year when used consistently and correctly ) from at least 7 days prior to vaccination until the end of the study or females who are permanently sterilized (at least 6 weeks post-sterilization).
7. Males who agree to apply effective contraception methods from day 0 through day 56.
8. Be willing to refrain from blood donation during the course of the study.
9. The subject is co-operative and available for the entire study.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria are met at screening or at day -1:

1. Prior receipt of a MERS vaccine or MVA immunizations.
2. Receipt of any vaccine in the 2 weeks prior to 1st trial vaccination (4 weeks for live vaccines) or planned receipt of any vaccine in the 3 weeks following the 2nd trial vaccination.
3. Known allergy to the components of the MVA-MERS-S vaccine product as eggs, chicken proteins, and gentamycin or history of life-threatening reactions to vaccine containing the same substances.
4. Participation in a clinical trial or use of an investigational product within 30 days or five times the half-life of the investigational drug -whichever is longer- prior to receiving the first dose within this study.
5. Evidence in the subject's medical history or in the medical examination that might influence either the safety of the subject or the absorption, distribution, metabolism or excretion of the investigational product under investigation.
6. Any positive result for human immunodeficiency virus (HIV)1/2 antibody, hepatitis C virus (HCV) antibody or hepatitis B surface antigen (HBsAg) testing.
7. Any confirmed or suspected immunosuppressive or immunodeficient condition, cytotoxic therapy in the previous 5 years, and/or diabetes.
8. Participants with inflammatory, infectious and neuroinflammatory underlying disease which could cause an expected impairment of the blood brain barrier such as meningitis, multiple sclerosis, epilepsy, or Alzheimer's disease.
9. Any chronic or active neurologic disorder, including migraines, seizures, and epilepsy, excluding a single febrile seizure as a child.
10. Known history of Guillain-Barré Syndrome.
11. Active malignancy or history of metastatic or hematologic malignancy.
12. Suspected or known alcohol and/or illicit drug abuse within the past 5 years.
13. Moderate or severe illness and/or fever >38°C within 1 week prior to vaccination.
14. Administration of immunoglobulins and/or any blood products within the 120 days preceding study entry or planned administration during the study period.
15. History of blood donation within 60 days of enrollment or plans to donate within the treatment phase (until the 2nd vaccination).
16. Receipt of chronic (defined as more than 14 days) immune suppressants or other immune-modifying drugs within 6 months of study inclusion (screening).

    * For corticosteroids, this will mean prednisone, or equivalent, greater than or equal to 0.5 mg/kg/day.
    * Intranasal and topical steroids are allowed.
17. Participants with skin lesions close to the injection site or active oral lesions will be excluded.
18. Thrombocytopenia, contraindicating intramuscular vaccination based on investigator's judgment.
19. Participants with a significant infection or known inflammation.
20. History of relevant cardiovascular disorders or evidence of hyper- (sitting blood pressure systolic >140 or diastolic >90 mmHg) or hypotension (sitting blood pressure systolic <90 or diastolic <40 mmHg) at screening.
21. Subjects who are known or suspected not to comply with the study directives.
22. Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marylyn M Addo, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- CTC North GmbH & Co. KG at the University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zaki AM, van Boheemen S, Bestebroer TM, Osterhaus AD, Fouchier RA. Isolation of a novel coronavirus from a man with pneumonia in Saudi Arabia. N Engl J Med. 2012 Nov 8;367(19):1814-20. doi: 10.1056/NEJMoa1211721. Epub 2012 Oct 17. PMID 23075143
- [Background] Memish ZA, Zumla AI, Al-Hakeem RF, Al-Rabeeah AA, Stephens GM. Family cluster of Middle East respiratory syndrome coronavirus infections. N Engl J Med. 2013 Jun 27;368(26):2487-94. doi: 10.1056/NEJMoa1303729. Epub 2013 May 29. PMID 23718156
- [Background] van Boheemen S, de Graaf M, Lauber C, Bestebroer TM, Raj VS, Zaki AM, Osterhaus AD, Haagmans BL, Gorbalenya AE, Snijder EJ, Fouchier RA. Genomic characterization of a newly discovered coronavirus associated with acute respiratory distress syndrome in humans. mBio. 2012 Nov 20;3(6):e00473-12. doi: 10.1128/mBio.00473-12. PMID 23170002
- [Background] Agnihothram S, Gopal R, Yount BL Jr, Donaldson EF, Menachery VD, Graham RL, Scobey TD, Gralinski LE, Denison MR, Zambon M, Baric RS. Evaluation of serologic and antigenic relationships between middle eastern respiratory syndrome coronavirus and other coronaviruses to develop vaccine platforms for the rapid response to emerging coronaviruses. J Infect Dis. 2014 Apr 1;209(7):995-1006. doi: 10.1093/infdis/jit609. Epub 2013 Nov 18. PMID 24253287
- [Background] Song F, Fux R, Provacia LB, Volz A, Eickmann M, Becker S, Osterhaus AD, Haagmans BL, Sutter G. Middle East respiratory syndrome coronavirus spike protein delivered by modified vaccinia virus Ankara efficiently induces virus-neutralizing antibodies. J Virol. 2013 Nov;87(21):11950-4. doi: 10.1128/JVI.01672-13. Epub 2013 Aug 28. PMID 23986586
- [Background] Sutter G, Moss B. Nonreplicating vaccinia vector efficiently expresses recombinant genes. Proc Natl Acad Sci U S A. 1992 Nov 15;89(22):10847-51. doi: 10.1073/pnas.89.22.10847. PMID 1438287
- [Background] Haagmans BL, van den Brand JM, Raj VS, Volz A, Wohlsein P, Smits SL, Schipper D, Bestebroer TM, Okba N, Fux R, Bensaid A, Solanes Foz D, Kuiken T, Baumgartner W, Segales J, Sutter G, Osterhaus AD. An orthopoxvirus-based vaccine reduces virus excretion after MERS-CoV infection in dromedary camels. Science. 2016 Jan 1;351(6268):77-81. doi: 10.1126/science.aad1283. Epub 2015 Dec 17. PMID 26678878
- [Derived] Weskamm LM, Fathi A, Raadsen MP, Mykytyn AZ, Koch T, Spohn M, Friedrich M; MVA-MERS-S Study Group; Haagmans BL, Becker S, Sutter G, Dahlke C, Addo MM. Persistence of MERS-CoV-spike-specific B cells and antibodies after late third immunization with the MVA-MERS-S vaccine. Cell Rep Med. 2022 Jul 19;3(7):100685. doi: 10.1016/j.xcrm.2022.100685. PMID 35858586
- [Derived] Fathi A, Dahlke C, Krahling V, Kupke A, Okba NMA, Raadsen MP, Heidepriem J, Muller MA, Paris G, Lassen S, Kluver M, Volz A, Koch T, Ly ML, Friedrich M, Fux R, Tscherne A, Kalodimou G, Schmiedel S, Corman VM, Hesterkamp T, Drosten C, Loeffler FF, Haagmans BL, Sutter G, Becker S, Addo MM. Increased neutralization and IgG epitope identification after MVA-MERS-S booster vaccination against Middle East respiratory syndrome. Nat Commun. 2022 Jul 19;13(1):4182. doi: 10.1038/s41467-022-31557-0. PMID 35853863
- [Derived] Koch T, Dahlke C, Fathi A, Kupke A, Krahling V, Okba NMA, Halwe S, Rohde C, Eickmann M, Volz A, Hesterkamp T, Jambrecina A, Borregaard S, Ly ML, Zinser ME, Bartels E, Poetsch JSH, Neumann R, Fux R, Schmiedel S, Lohse AW, Haagmans BL, Sutter G, Becker S, Addo MM. Safety and immunogenicity of a modified vaccinia virus Ankara vector vaccine candidate for Middle East respiratory syndrome: an open-label, phase 1 trial. Lancet Infect Dis. 2020 Jul;20(7):827-838. doi: 10.1016/S1473-3099(20)30248-6. Epub 2020 Apr 21. PMID 32325037
- See also: Middle East respiratory syndrome coronavirus situation updates — http://www.who.int/emergencies/mers-cov/en/

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccination With 10^7 PFU MVA-MERS-S; Vaccination With 10^8 PFU MVA-MERS-S: Vaccinations occur on days 0 and 28
  A subgroup will additionally receive a late booster immunization with 10^8 PFU MVA-MERS-S 12 months (+/- 4 months) after prime immunization.
  vaccine candidate MVA-MERS-S: vaccination with MVA-MERS-S in two escalating dose regimes
Period: Overall Study
Arm/Group | Vaccination With 10^7 PFU MVA-MERS-S | Vaccination With 10^8 PFU MVA-MERS-S
Started | 14 | 12
Received Late Booster Immunization | 3 | 7
Completed | 12 (A subgroup received an additional booster of 1x10^8 PFU MVA-MERS-S 12 (+/-4) months after prime.) | 11 (A subgroup received an additional booster of 1x10^8 PFU MVA-MERS-S 12 (+/-4) months after prime.)
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccination With 10^7 PFU MVA-MERS-S | Vaccination With 10^8 PFU MVA-MERS-S | Total
Number analyzed (Participants) | 14 | 12 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 12 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 4 | 2 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 13 | 11 | 24
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 14 | 12 | 26
BMI (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 23.6 (2.5) | 23.5 (3.7) | 23.6 (3.0)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Experiencing Solicited Local or Systemic Reactogenicity as Defined by the Study Protocol
Description: The solicited local adverse events for this study include:
  Swelling, erythema, induration, hematoma and pain at site of injection
  The solicited systemic adverse events for this study include:
  * Fever
  * Chills
  * Myalgia (described to the subject as generalized muscle aches)
  * Arthralgia (described to the subject as generalized joint aches)
  * Fatigue/Malaise
  * Headache
  * Gastrointestinal symptoms
  The reactogenicity (adverse events) will be assessed via a trained physician taking into account a patient diary. The severity of the adverse event will be measured as specified in the study protocol (grade 0=none, grade 1=mild, grade 2=moderate, grade 3=severe). The adverse event will furthermore be categorized in related vs. not related.
Time Frame: 14 days after each vaccination
Measure: Count of Participants; unit: Participants
Groups:
- Vaccination With 10^7 PFU MVA-MERS-S; Vaccination With 10^8 PFU MVA-MERS-S: Vaccinations occur on days 0 and 28.
  A subgroup will additionally receive a late booster immunization with 10^8 PFU MVA-MERS-S 12 months (+/- 4 months) after prime immunization.
Arm/Group | Vaccination With 10^7 PFU MVA-MERS-S | Vaccination With 10^8 PFU MVA-MERS-S
Number analyzed (Participants) | 14 | 12
Participants | 10 | 10

2. Primary Outcome: Percentage of Participants Who Experienced an Unsolicited Adverse Event
Description: The unsolicited adverse events will be assessed via a trained physician taking into account a patient diary. The severity of the adverse event will be measured as specified in the study protocol (grade 0=none, grade 1=mild, grade 2=moderate, grade 3=severe). The adverse event will furthermore be categorized in related vs. not related.
Time Frame: 28 days after each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination With 10^7 PFU MVA-MERS-S | Vaccination With 10^8 PFU MVA-MERS-S
Number analyzed (Participants) | 14 | 12
Participants | 5 | 8

3. Primary Outcome: Change of Mean C-reactive Protein (CRP) Levels (Measured in [mg/l]) From Baseline (Day -1 ) as Compared to the End of the Study (D180)
Description: The safety laboratory measures include:
  - Clinical Chemistry: CRP in miligrams per liter [mg/l]
Time Frame: Throughout the study up to conclusion
Population: All participants were included in the safety analysis.
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Vaccination With 10^7 PFU MVA-MERS-S | Vaccination With 10^8 PFU MVA-MERS-S
Number analyzed (Participants) | 14 | 12
mg/l | 0 (0.3) | -1 (3)

4. Primary Outcome: Change of Mean White Blood Cell (WBC) Counts (Measured in [Billion Cells/L]) From Baseline (Day -1) as Compared to the End of the Study (D180)
Description: The safety laboratory measures include Hematology: WBC count in billions per liter [billion cells/L]
Time Frame: Throughout the study up to conclusion
Measure: Mean (Standard Deviation); unit: Billion Cells/L
Arm/Group | Vaccination With 10^7 PFU MVA-MERS-S | Vaccination With 10^8 PFU MVA-MERS-S
Number analyzed (Participants) | 14 | 12
Billion Cells/L | -1.8 (1.44) | -1.0 (1.92)

5. Primary Outcome: Percentage of Participants Experiencing a Serious Adverse Event up to Day 180 (Study Completion)
Description: Serious adverse events are defined as any untoward medical occurrence (whether considered to be related to investigational medicinal product or not) that at any dose:
  * results in death
  * is life-threatening
  * requires inpatient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * is a congenital abnormality/birth defect
  * is an Important Medical Event, i.e., an event that may jeopardize the subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: Throughout the study up to conclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination With 10^7 PFU MVA-MERS-S | Vaccination With 10^8 PFU MVA-MERS-S
Number analyzed (Participants) | 14 | 12
Participants | 0 | 0

6. Secondary Outcome: Immunogenicity: Number of Participants Who Seroconverted Throughout the Study (up to Study Completion at Day 180)
Description: Humoral immunity: The magnitude of MVA-MERS-S antibody responses as assessed by neutralization assay and ELISA.
Time Frame: Throughout the study up to conclusion
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccination With 10^7 PFU MVA-MERS-S | Vaccination With 10^8 PFU MVA-MERS-S
Number analyzed (Participants) | 12 | 11
Participants | 8 | 10

ADVERSE EVENTS:
Time Frame: Solicited AE: 14 days after each vaccination Unsolicited AE: 28 days after each vaccination SAE: Throughout the study (180 days). In case of participation in the follow-up booster immunization 12 months (+/-4 months after prime vaccination) additional 28-day follow-up time after booster vaccination.
Description: Participants filled out a participant diary, which was assessed on study visits (Day 1, 3, 7, 14, 28 after vaccination).
Arm/Group | Vaccination With 10^7 PFU MVA-MERS-S | Vaccination With 10^8 PFU MVA-MERS-S
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 10/14 | 10/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccination With 10^7 PFU MVA-MERS-S (N=14) | Vaccination With 10^8 PFU MVA-MERS-S (N=12)
Local reactogenicity (Skin and subcutaneous tissue disorders) | 8 | 10 — The Analysis of Adverse Events of the late booster subgroup are part of the exploratory objectives of the study, not part of the statistical analysis plan and are therefore not included here.
Fatigue and Malaise (General disorders) | 10 | 7
Gastrointestinal Symptoms (Gastrointestinal disorders) | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Headache (Nervous system disorders) | 7 | 9
Other systemic unsolicited (General disorders) | 1 | 1
Fever/Chills (Immune system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT03615911/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03615911/SAP_001.pdf